CLINICAL TRIAL: NCT06784960
Title: A Cluster Randomized Controlled Trial Testing Communication Strategies to Increase HPV Vaccination Intention: a Survey Experiment
Brief Title: Communication Strategies to Increase HPV Vaccination Intention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Florence Momplaisir, MD, Associate Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 856892
Record Dates: First submitted 2024-12-12; First posted 2025-01-20 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Papilloma Viral Infection; Vaccine Hesitancy; Communication
MeSH Terms: conditions — Papillomavirus Infections; Vaccination Hesitancy; Communication

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Theory-Based Message Condition 1 (Experimental)
  Interventions: Behavioral: Messages
- Theory-Based Message Condition 2 (Experimental)
  Interventions: Behavioral: Messages
- Theory-Based Message Condition 3 (Experimental)
  Interventions: Behavioral: Messages
- Theory-Based Message Condition 4 (Experimental)
  Interventions: Behavioral: Messages
- Theory-Based Message Condition 5 (Experimental)
  Interventions: Behavioral: Messages
- Theory-Based Message Condition 6 (Active Comparator)
  Interventions: Behavioral: Messages

INTERVENTIONS:
Behavioral: Messages — We will randomly assign participants in equal numbers to one of five theory-based HPV vaccine message conditions or an attention-matched control arm.

SUMMARY:
This research aims to identify communication strategies to improve the uptake of vaccines using an experimental design, focusing on the Human Papillomavirus (HPV) vaccine, which is highly effective in preventing HPV-related cancers. However, low HPV vaccination rates among adults remain a significant public health challenge. Although randomized controlled trials (RCTs) have demonstrated that interventions can increase vaccine uptake in children, few RCTs have been conducted on adults. To address this gap, a multidisciplinary investigative team with expertise in communication, medicine, nursing, and behavior-change intervention research, and a history of extensive collaboration, will conduct a survey experiment on a national sample of over 3,689 adults to identify the most promising theory-based messages to strengthen HPV vaccine intentions.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old

Exclusion Criteria:

* Under 18 and over 45 years old
* Received HPV vaccine or unsure about receipt

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3689 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Intention to Vaccinate | Immediately after the intervention
  Validated 3-item likert scale assessing HPV vaccination intention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No